CLINICAL TRIAL: NCT04597801
Title: Comparison of Fluorescein-INtra-VItal Microscopy Versus Conventional Frozen Section Diagnosis for intraOperative Histopathological Evaluation (INVIVO)
Brief Title: Comparison of Fluorescein-INtra-VItal Microscopy Versus Conventional Frozen Section Diagnosis for intraOperative Histopathological Evaluation
Acronym: INVIVO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INV-GEM-0200-I
Record Dates: First submitted 2020-09-14; First posted 2020-10-22 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-04

CONDITIONS: Intracranial Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — methylacetylene; Fluorescein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fluorescein sodium (Experimental): A single dose of fluorescein sodium is applied before brain tumor resection. 20-40 minutes prior to the planned tumor resection, a bolus of 5 mg per kg body weight is administered intravenously, staining tumor tissue with fluorescent dye to visualize tumor cells.
  Interventions: Drug: Alcon

INTERVENTIONS:
Drug: Alcon — Fluorescein sodium is administered intravenously with a bolus injection of 5 mg per kg of bodyweight 20-40 minutes prior to the planned tumor resection.
  Other Names: Fluorescein sodium

SUMMARY:
With the appliance of the in-vivo microscopy after Fluorescein staining, the investigators hypothesize that the preliminary in-vivo histopathological diagnostic accuracy is not inferior to conventional frozen section analysis accuracy when using the final histopathological result as gold standard.

DETAILED DESCRIPTION:
In neurosurgery, intraoperative histopathological frozen section analysis (cryosection) offers a crucial tool for the rapid assessment of tumor entity and dignity and the creation of tumor-free resection margins. The method, however, remains unreliable and time-consuming, sometimes prolonging surgical times and demonstrating diagnostic accuracy for frozen section in glioma ranging from 78.4% to 95% in comparison to the final histopathology, depending on the technique used.2,3 To combat these shortcomings, another promising adjunct was developed in the form of intraoperative dye-dependent in-vivo microscopy, for which there has been little scientific evidence so far, with only a few recent studies exploring its utility, safety and general applicability. The theoretical idea of the technique in principle is to allow for histopathological assessment of tumor tissue in-vivo without the need for time-consuming fixation and transport of resected tissue biopsies, aiming for a so-called in-situ digital biopsy and thereby substantially improving operative precision and surgical times. It stands to reason that the benefit in visualization provided by fluorescein staining may further be driven through in-vivo microscopy. Altogether, with the use of fluorescein sodium in in-vivo microscopy, the operating surgeon may in the future inspect supposedly malignant fluorescent tissue first-hand, evaluate it for tumorous cells in real-time and adjust their resection strategy in a far more immediate fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Signed informed consent
3. Suspected intracranial tumor revealed by cranial magnetic resonance imaging (according to clinical routine) scheduled for resection with intraoperative frozen section evaluation

Exclusion Criteria:

1. Known allergic or suspected allergic reactions to fluorescein sodium
2. Liver disease, CHILD B or C
3. Patients under medication with beta-blockers, digoxin, chinidin and probenecid as well as inhibitors of glucuronidation, such as immunosuppressants, when the medication must not be discontinued perioperatively
4. Patients with relevant congenital limitations of glucuronidation performance (e.g. Rotor syndrome, Gilbert-Meulengracht syndrome, Crigler-Najjar syndrome)
5. Patients with terminal renal failure requiring hemodialysis
6. Inability to provide informed consent
7. Pregnancy (incl. positive pregnancy test)
8. Women of childbearing age must be non-lactating and surgically sterile or using a highly effective method of birth control and have a negative pregnancy test. Acceptable methods of birth control with a low failure rate (i.e. less than 1% per year) when used consistently and correct are such as implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomized partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Significance: The diagnostic accuracies of the individual methods used for preliminary intraoperative histopathological diagnosis (D1:fluorescein sodium with in-vivo microscopy versus D2: preliminary frozen section assessment) | 14 days
  The primary objective of the clinical trial is to compare the significance of intravenously applied fluorescein as staining agent for assessment of brain tissue texture via in-vivo confocal microscopy with the conventional intraoperative histological frozen section analysis of identical brain tissue samples in the same patient. Both methods will be compared in terms of their accuracy using the standard of practice, the final pathological diagnosis (immunochemistry/molecular pathology).

SECONDARY OUTCOMES:
Incidence of adverse events during surgery and until end of follow-up period (Safety Assessment) | 24 days
  To assess the safety of the Investigational Medicinal Product (IMP) as staining agent for in-vivo confocal microscopy by documentation of adverse events during surgery and until end of follow-up period.
Analysis of surgical time span (comparison of the time span to conduct the assessment of brain tissue texture with fluorescein intervention with the time span to conduct assessment of conventional intraoperative frozen section intervention. | 14 days
  Analysis of surgical time span: comparison of the time span to conduct the assessment of brain tissue texture with fluorescein intervention with the time span to conduct assessment of conventional intraoperative frozen section intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jens PD Gempt, MD, Study Chair — Technische Universität München, Klinik und Poliklinik für Neurochirurgie
Locations (3):
- Germany (3):
  - Universitätsklinikum Mannheim, Mannheim
  - Technische Universität München, Klinik und Poliklinik für Neurochirurgie, München
  - Universitätsklinikum Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No
IPDs will not be shared